CLINICAL TRIAL: NCT00313807
Title: CoNTRST - Contrast Nephropathy and Travasol for Renal Safety Trial: Intravenous Amino Acid Infusion for the Prevention of Contrast-mediated Acute Renal Failure Following Coronary Catheterization
Brief Title: Study of Intravenous Amino Acid Infusion to Prevent Contrast Dye Mediated Renal Damage
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandoned due to lack of recruitment Oct 2006
Sponsor: Queen's University (Other)
Responsible Party: Dr Karen E. Yeates, Department of Medicine Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: contrst2006
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Contrast Nephropathy; Renal Failure
Keywords: contrast nephropathy; renal failure; Travasol
MeSH Terms: conditions — Renal Insufficiency | interventions — Amino Acids; Parenteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intravenous saline infusion plus amino acid infusion
  Interventions: Drug: Amino Acid
- 2 (Placebo Comparator): Intravenous saline infusion plus placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amino Acid — 7% amino acid infusion
  Other Names: Parenteral nutrition
  Arms: 1
Drug: Placebo — 0.9% Saline Infusion
  Other Names: Normal Saline Infusion
  Arms: 2

SUMMARY:
Exposure to radiographic contrast dye during coronary angiography is well known to cause either transient decreases in renal function or acute renal failure. Although the overall incidence is low, acute renal failure occurs most frequently in patients with both diabetes and chronic renal failure where the average reported incidence is upwards of 20%. The etiology of contrast-induced nephropathy is related to acute decline in renal blood flow following dye exposure resulting in ischemic injury at the level of the medulla. The development of acute renal failure following radiocontrast dye administration is significant because it contributes to morbidity and mortality in patients at risk.

The administration of amino acids, either through intravenous infusion or a protein meal, results in a substantial increase in renal plasma flow (RPF) and glomerular filtration rate (GFR). In both healthy subjects and in those with chronic renal failure, an amino acid infusion produces a 20% rise in GFR and effective RPF.

We hypothesize that the 20% rise in effective RPF and GFR following an amino acid infusion will counteract the radiocontrast dye-induced vasoconstriction and reduce the renal toxicity of contrast medium in a group of high-risk patients.

DETAILED DESCRIPTION:
Exposure to radiographic contrast dye during coronary angiography is well known to cause either transient decreases in renal function or acute renal failure.

Retrospective studies have confirmed that at least 60% of contrast-associated nephropathy occurs in subjects with chronic renal failure. The incidence approaches 20% in those with a baseline creatinine greater than 198.2 μmol per liter (2.25 mg/dL). Diabetes, in the absence of renal insufficiency, does not appear to confer added risk; however diabetic patients with chronic renal failure are at highest risk. It is particularly this group that develops oliguric renal failure requiring temporary or permanent renal replacement therapy. In diabetic patients with mild to moderate renal failure, the incidence of contrast-associated nephropathy has been reported to be between 9% and 40% however a greater then 50% incidence has been noted in diabetic patients with more severely impaired renal function.

It is hypothesized that the renal toxicity of contrast medium is related to local vasoconstriction. We hypothesize that the protein-stimulated rise in effective RPF and GFR might counteract this intrarenal vasoconstriction and reduce the toxicity of contrast medium in high-risk patients with diabetes. We propose that an infusion of amino acids prior to the administration of contrast dye, will increase renal plasma flow and glomerular filtration rate by approximately 20% and hasten excretion of the contrast agent thereby protecting high-risk patients from contrast nephropathy.

This is a double-blind, randomized, placebo-controlled trial evaluating the effectiveness of an amino-acid infusion in addition to usual therapy (intravenous normal saline infusion) for the prevention of renal dysfunction following angiographic dye administration during coronary angiography in a high risk group of patients with chronic renal insufficiency.

Comparison: Primary and secondary outcomes in patients receiving intravenous amino acid infusion compared to placebo group receiving intravenous normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Greater then 18 years of age
* Referral for coronary angiography
* Type 1 or type 2 diabetic requiring insulin or oral hypoglycemic agents
* Stable serum creatinine concentration (140 to 300 μmol per liter for men or 125 to 300 μmol per liter for women or a creatinine clearance not greater than 60 ml/min (as calculated by Cockcroft-Gault equation)
* Non diabetic subjects with a stable serum creatinine concentration of 160 to 300 µmol per liter for men and 140 to 300 µmol per liter for women.
* Stable renal function defined as no documented rise or fall in serum creatinine by more then 44 umol/L in the preceding 2 weeks

Exclusion Criteria:

* Refusal or inability to give consent
* Pregnant
* Non-elective coronary angiography
* Recent administration (within 21 days) of iodinated intravenous contrast dye
* Recent administration (within 21 days) of non-steroidal anti-inflammatory drugs (excluding aspirin), aminoglycoside antibiotics or chemotherapeutic agents
* Severe/unstable diabetics requiring emergency room or inpatient therapy in the previous 21 days
* Compensated or decompensated hepatic failure
* Renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Study Completion 2008-09

PRIMARY OUTCOMES:
to assess if the infusion of amino acids will help prevent kidney damage that can occur when angiographic dye is used to perform a cardiac catheterization | Day 0 to Day 7

SECONDARY OUTCOMES:
the serum cystatin C level at 24 hours post procedure and 72 hours post procedure | Day 0 to Day 3
the number of patients with a peak increase in serum creatinine concentration of at least 44.1 umol/L between day 0 and day 3 (72 hours) | Day 0 to Day 3
the number of patients with a peak increase in serum creatinine concentration of at least 88.4 μmol per liter between day 0 and day 3 (72 hours) post-catheterization | Day 0 to Day 3
development of heart failure or myocardial infarction within 7 days | 7 days
need for renal replacement therapy | 7days
death at 48 hours, 7 days, or 14 days post-catheterization | 14 days
number of hospital days after catheterization | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Yeates, MD MPH, Principal Investigator — Assistant Professor, Queen's University - Division of Nephrology, Department of Medicine